CLINICAL TRIAL: NCT04966793
Title: Microbial Colonization Distribution and Adaptive Evolution of Lower Respiratory Tract in Bronchiectasia Patients.
Brief Title: Microbial Colonization Distribution and Adaptive Evolution of Lower Respiratory Tract in Bronchiectasis Patients.
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); Xuanwu Hospital, Beijing (Other); Nanjing Jiangning Hospital (Unknown); Tongji Hospital (Other); Huadong Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Chest Hospital, Capital Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Shandong Public Health Clinical Center (Other Government); The First Medical Center of Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-066
Record Dates: First submitted 2021-06-07; First posted 2021-07-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-06

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Microbiology
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bronchiectasis patients group: Bronchiectasis patients group: Sputum specimens from bronchiectasis patients aged 18 to 79 years old .
- Healthy control group: Healthy control group: Sputum specimens from healthy people.

SUMMARY:
Qualified sputum samples from bronchiectasis patients were collected regularly every month for three consecutive years to analyze the microbiome changes of lower respiratory tract of bronchiectasis patients by metagenomic sequencing. Pseudomonas aeruginosa was isolated and the whole genome was sequenced to analyze the adaptive evolution，including virulence, quorum sensing and drug resistance under host pressure. The aim of the study is to clarify the rule of microflora colonization distribution and adaptive evolution in the lower respiratory tract of patients with bronchiectasis, to predict the acute attack and prognosis of patients with microbiome changes, and to find more new prevention and treatment methods by adjusting the microbiome of the lower respiratory tract.

DETAILED DESCRIPTION:
Bronchiectasis is an abnormal, permanent dilatation of the bronchi, which presents as cough, expectoration and recurrent pulmonary infections. Epidemiological survey researchs have found that the number of bronchiectasis has increased rather than decreased in the last decades. Asia has the highest prevalence of bronchiectasis, with 1,200 cases in every 100,000 people over the age of 40 in China, and this rate can be seriously underestimated due to difficulties in identifying COPD. The mortality rate of bronchiectasis patients is more than twice that of the general population, placing an increasing burden on global health care systems. Chronic infection in bronchiectasis is common and had a big influence on prognosis. Pseudomonas aeruginosa is considered to be the most common colonization bacterium. At present, the mechanism of bronchiectasis and its relationship with lower respiratory tract infection have not been fully elucidated. Therefore, it is important to have an in-depth understanding of the colonization distribution and adaptive evolution of the microbiome in the lower respiratory tract, to predict the acute attack and prognosis with the application of microbiome changes, and to find more new and effective prevention and treatment methods by regulating the microbiome in the lower respiratory tract. Qualified sputum specimens from bronchiectasis patients were collected regularly every month for three consecutive years. Metagenomic sequencing was used to analyze the microbiome changes of lower respiratory tract in these patients. Pseudomonas aeruginosa was isolated and the whole genome was sequenced to analyze the adaptive evolution of its virulence, group sensitivity and drug resistance under host pressure.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiectasis patients in clinically stable period;
* Two or more chest infections in the previous year;
* Chest CT confirmed bronchiectasis (bronchial to arterial ratio >1).
* Chronic colonization of pseudomonas aeruginosa and was clinically stable in 6 months prior to the study.

Exclusion Criteria:

* deterioration of illness (defined as at least 24 hours of three or more of the following symptoms: increased cough, increased sputum volume, purulent sputum, hemoptysis, increased dyspnea, increased wheezing, fever ((≥38°C) or discomfort, the attending physician agrees that antibiotic treatment is required);
* current smokers, or former smokers who have stopped smoking less than 1 year ago, have a history of more than 15 packets of age, or CT showed as emphysema;
* cystic fibrosis patients;
* active allergic bronchopulmonary aspergillosis;
* active tuberculosis patients;
* patients with poor asthma control;
* pregnant or breastfeeding women.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bronchiectasis patients aged 18 to 79.
Sampling Method: Probability Sample
Enrollment: 1850 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline SNP of PA population in sputum samples | once per 3 month for 3 years
  To assess the SNP changes of PA population in sputum samples compared with PAO1 wildtype
Species richness and antibiotic suscepibility change from baseline in sputum samples | once per 3 month for 3 years
  To assess the species richness and antibiotic suscepibility change from baseline in sputum samples

SECONDARY OUTCOMES:
pulmonary function | once per year for 3 years
  To assess the lung functon change
chest CT | once per year for 3 years
  To assess the severity of lung lesions
BSI scores | once per year for 3 years
  To assess the severity index of bronchiectasis.
E-FACED scores | once per year for 3 years
  To assess the severity index of bronchiectasis.
SGRQ questionnaire | once per year for 3 years
  To assess the impaired health and quality of life of patients with respiratory diseases

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China